CLINICAL TRIAL: NCT00003145
Title: Induction of Mixed Hematopoietic Chimerism Using Fludarabine, Low Dose TBI , PBSC Infusion and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil to be Followed by Donor Lymphocyte Infusion In Patients With Chronic Myeloid Leukemia in Chronic and Accelerated Phases: A Multi-center Study
Brief Title: Fludarabine Phosphate, Low-Dose Total-Body Irradiation, and Peripheral Blood Stem Cell Transplant Followed by Donor Lymphocyte Infusion in Treating Older Patients With Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1209.00; NCI-2012-00579 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1209.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Accelerated Phase of Disease; Childhood Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase of Disease; Recurrent Disease
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Recurrence | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, TBI, PBSCT, DLI) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID or IV BID or TID on days -3 to 56 with taper to day 77 or 180, and mycophenolate mofetil PO or IV BID on days 0-27.
  DLI: At least 2 weeks after completion of immunosuppression, patients with > 5% donor CD3+ T cells and no evidence of GVHD receive donor lymphocytes IV over 30 minutes. Patients may receive up to 3 DLIs at increasing cell doses in the absence of GVHD.
  Interventions: Drug: Fludarabine Phosphate; Radiation: Total-Body Irradiation; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Cyclosporine; Drug: Mycophenolate Mofetil; Biological: Therapeutic Allogeneic Lymphocytes; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole-Body Irradiation
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; CsA; Neoral; OL 27-400; Sandimmun
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Biological: Therapeutic Allogeneic Lymphocytes — Given IV
  Other Names: Allogeneic Lymphocytes; ALLOLYMPH; Tumor-Derived Lymphocyte
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies fludarabine phosphate, low-dose total-body irradiation, and peripheral blood stem cell transplant followed by donor lymphocyte infusion in treating older patients with chronic myeloid leukemia. Giving chemotherapy and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect). Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if mixed hematopoietic chimerism can be safely established using a non-myeloablative conditioning regimen in patients > 65 years of age with chronic myeloid leukemia (CML) in chronic or accelerated phase who have human leukocyte antigen (HLA) identical related donors.

II. To determine if mixed chimerism, established with non-myeloablative conditioning regimens, can be converted to full donor hematopoietic chimerism by infusions of donor lymphocytes (DLI), and thereby produce an immunologic cure of the malignancy.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo low-dose total-body irradiation (TBI) on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) or IV BID or thrice daily (TID) on days -3 to 56 with taper to day 77 or 180, and mycophenolate mofetil PO or IV BID on days 0-27.

DLI: At least 2 weeks after completion of immunosuppression, patients with > 5% donor cluster of differentiation (CD)3+ T cells and no evidence of graft-versus-host disease (GVHD) receive donor lymphocytes IV over 30 minutes. Patients may receive up to 3 DLIs at increasing cell doses in the absence of GVHD.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia chromosome positive (Ph+) CML in first and second chronic and first accelerated phases
* Patients =< 65 years old who are at high risk of regimen related toxicity through pre-existing chronic disease affecting liver, lungs, and/or heart, or others who wish to be treated on this protocol, will be considered on a case-by-case basis; transplants should be approved for these inclusion criteria by both the participating institutions' patient review committees such as the Patient Care Conference (PCC) at the Fred Hutchinson Cancer Research Center (FHCRC) and by the principal investigators at the collaborating centers; patients =< 65 years of age who have received previous high-dose transplantation do not require patient review committee approvals; all children < 12 years must be discussed with the FHCRC principal investigator (PI) (Brenda Sandmaier, MD 206-667-4961) prior to registration
* HLA genotypically identical related donor willing to undergo leukapheresis initially for collection of peripheral blood stem cell (PBSC) and subsequently for collection of peripheral blood mononuclear cell (PBMC)
* Patients treated with alpha interferon must have discontinued drug at least 1 month prior to transplant
* DONOR: HLA genotypically identical family member (excluding identical twins)
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)

Exclusion Criteria:

* Patients who are human immunodeficiency virus positive (HIV+)
* GROUP 1: (PATIENTS AGED > 65 AND < 75 YEARS)
* Patients unwilling to use contraceptive techniques during and for 12 months following treatment
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with CML
* Patients in an interferon induced complete or partial cytogenetic remission
* Organ dysfunction:

  * Patients with renal failure are eligible, however patients with renal compromise (Serum creatinine greater than 2.0) will likely have further compromise in renal function and may require hemodialysis (which may be permanent) due to the need to maintain adequate serum cyclosporine levels
  * Cardiac ejection fraction < 40%; ejection fraction is required if the patient has a history of anthracyclines or history of cardiac disease
  * Diffusing capacity of the lung for carbon monoxide (DLCO) < 50% of predicted
  * Liver function tests including total bilirubin, serum glutamic pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) > 2x the upper limit of normal unless proven to be due to the malignancy
  * Karnofsky score < 70
* Patients with poorly controlled hypertension
* GROUP 2 (PATIENTS AGED =< 65)
* Patients who are HIV+
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with CML
* Females who are pregnant
* Patients unwilling to use contraceptive techniques during and for 12 months following treatment
* Patients in an interferon induced complete or partial cytogenetic remission
* Organ dysfunction:

  * Patients with renal failure are eligible, however patients with renal compromise (Serum creatinine greater than 2.0) will likely have further compromise in renal function and may require hemodialysis (which may be permanent) due to the need to maintain adequate serum cyclosporine levels
  * Cardiac ejection fraction < 40% or a history of congestive heart failure; ejection fraction is required if the patient has a history of anthracyclines or history of cardiac disease
  * Severe defects in pulmonary function testing as defined by the pulmonary consultant (defects are currently categorized as mild, moderate and severe) or receiving supplementary continuous oxygen; DLCO < 50% of predicted
  * Liver function tests: total bilirubin > 2x the upper limit of normal, SGPT and SGOT 4x the upper limit of normal
  * Karnofsky score < 50
* Patients with poorly controlled hypertension
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1997-08; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Safety of establishing mixed chimerism using this non-lethal conditioning regimen, in terms of development of GVHD, myelosuppression, infections, and treatment-related mortality | Within the first 65 days
  All unexpected toxicities will be summarized and reported.
Proportion of patients who successfully establish mixed chimerism (evidence of donor engraftment) and the proportion who convert to full donor chimeras among those who were mixed | Day 28
  Estimated and corresponding confidence intervals presented. Mixed chimerism is detection of donor T cells (CD3+) and granulocytes (CD33+), as proportion of total T cell and granulocyte population of > 5% and < 95% in peripheral blood. Full donor chimerism is > 95% donor CD3+ T cells. Increasing donor chimerism is absolute increase of 20% of CD3+ T cells over chimerism evaluation of previous month. Decreasing donor chimerism is absolute decrease of 20% of CD3+ T cell chimerism over previous month. Low donor chimerism is < 40% CD3+ T cells after HSCT.
Proportion of patients who successfully establish mixed chimerism (evidence of donor engraftment) and the proportion who convert to full donor chimeras among those who were mixed | Day 56
  Estimated and corresponding confidence intervals presented. Mixed chimerism is detection of donor T cells (CD3+) and granulocytes (CD33+), as proportion of total T cell and granulocyte population of > 5% and < 95% in peripheral blood. Full donor chimerism is > 95% donor CD3+ T cells. Increasing donor chimerism is absolute increase of 20% of CD3+ T cells over chimerism evaluation of previous month. Decreasing donor chimerism is absolute decrease of 20% of CD3+ T cell chimerism over previous month. Low donor chimerism is < 40% CD3+ T cells after HSCT.

SECONDARY OUTCOMES:
Proportion of patients experiencing a complete antileukemic response | At 12 weeks after the final DLI
  Reported in a descriptive manner and confidence intervals will be presented for all estimates.
Proportion of patients experiencing GVHD | Until day 90 after the last DLI
  Reported in a descriptive manner and confidence intervals will be presented for all estimates.
Proportion of patients experiencing non-relapse mortality | Within 65 days of transplant
  Reported in a descriptive manner and confidence intervals will be presented for all estimates.
Incidence of myelosuppression after initial PBSC infusion | Until 2 months post-transplant
  Defined as absolute neutrophil count [ANC] < 500 for > 2 days, platelets < 20,000 for > 2 days.
Incidence of aplasia after DLI | Until 2 months post-transplant
Incidence of grades 2-4 acute GVHD after DLI | Until day 90 after the last DLI
Incidence of grades 2-4 acute GVHD after PBSC infusion | Until day 90 after the last DLI
Incidence of grade chronic extensive GVHD after DLI | At 1 year
Dose of CD3+ cells required to convert mixed to full lymphoid chimeras | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (8):
- United States (6):
  - City of Hope Medical Center, Duarte, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - University of Colorado, Denver, Colorado
  - Baylor University Medical Center, Dallas, Texas
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- Universitaet Leipzig, Leipzig, Germany
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241